CLINICAL TRIAL: NCT07321197
Title: Template Lymph Node Dissection for Tumor Control in High-Risk Renal Cell Carcinoma: A Prospective, Open-Label, Multicenter, Randomized Controlled Trial
Brief Title: Radical Nephrectomy With vs Without Template Lymph Node Dissection in High-Risk Renal Cell Carcinoma (T-LND RCC): A Randomized Clinical Trial
Acronym: RECLND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Tianjin Third Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLND-RCC
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer)
Keywords: Template Lymph Node Dissection; High-Risk Neoplasm; Randomized Controlled Trial; Surgical Oncology
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Template Lymph Node Dissection (Experimental): Patients randomized to this arm will undergo radical nephrectomy (which may be performed via open, laparoscopic, or robot-assisted approach based on the surgeon's expertise) combined with a standardized template lymph node dissection.
  The template lymph node dissection is defined as follows:
  For Left-sided Tumors: Removal of lymphatic tissue anterior and lateral to the abdominal aorta, extending from the diaphragmatic crus superiorly to the aortic bifurcation inferiorly, including the renal hilar lymph tissue.
  For Right-sided Tumors: Removal of lymphatic tissue surrounding the inferior vena cava and in the interaortocaval space, extending from the liver edge of the vena cava superiorly to the iliac vein bifurcation inferiorly, including the renal hilar lymph tissue.
  Interventions: Procedure: Template Lymph Node Dissection
- Selective Lymph Node Resection (Active Comparator): Patients randomized to this arm will undergo radical nephrectomy (which may be performed via open, laparoscopic, or robot-assisted approach). In this arm, only lymph nodes that are identified as >1 cm in the short axis on preoperative cross-sectional imaging (CT/MRI) OR are grossly enlarged and suspicious during the surgeon's intraoperative assessment will be resected. If no such nodes are identified preoperatively or intraoperatively, no formal lymph node dissection is performed.
  Interventions: Procedure: Selective Lymph Node Resection

INTERVENTIONS:
Procedure: Template Lymph Node Dissection — A standardized surgical procedure to remove lymph nodes within defined anatomical boundaries during radical nephrectomy for kidney cancer. For left-sided tumors, this includes tissue anterior and lateral to the aorta from the diaphragmatic crus to the aortic bifurcation. For right-sided tumors, it includes tissue around the vena cava and between the vena cava and aorta from the liver edge to the iliac bifurcation. The renal hilar lymph tissue is always included.
  Arms: Template Lymph Node Dissection
Procedure: Selective Lymph Node Resection — A surgical approach during radical nephrectomy for kidney cancer where lymph nodes are removed only if they meet specific criteria: being larger than 1 cm on preoperative CT/MRI scans, or appearing grossly enlarged and suspicious to the surgeon during the operation. If no such nodes are identified, no lymph node dissection is performed.
  Arms: Selective Lymph Node Resection

SUMMARY:
The goal of this clinical trial is to learn if a more thorough lymph node removal surgery, called "Template Lymph Node Dissection," can help prevent cancer from returning and help patients live longer, compared to removing only a few enlarged lymph nodes, in patients with high-risk kidney cancer. The main questions it aims to answer are:

Do patients who receive template lymph node dissection live longer without their cancer returning (Disease-Free Survival)? Do patients who receive template lymph node dissection live longer overall (Overall Survival)? Is the more extensive lymph node surgery as safe as the limited surgery? Researchers will compare the Template Lymph Node Dissection group to the Limited Node Resection group to see the effects on cancer control and safety.

Participants will:

Be randomly assigned to one of the two surgical groups. Undergo surgery to remove their kidney and the assigned lymph nodes. Attend regular follow-up visits with imaging scans (like CT or MRI) for the first 5 years after surgery to monitor if the cancer returns.

Be followed for their overall survival status for up to 10 years.

DETAILED DESCRIPTION:
Research Background:

Renal cell carcinoma (RCC) remains a significant urological malignancy with rising global incidence. Radical nephrectomy (RN) is the standard curative treatment for localized disease. The therapeutic value of lymph node dissection (LND) in RCC, however, remains controversial. The EORTC 30881 trial demonstrated no survival benefit for RN with LND in clinically node-negative (cN0) patients, leading to its omission in contemporary guidelines. However, this trial predominantly included low-risk patients with a low incidence of pathological nodal involvement (4.0%), rendering it underpowered to evaluate LND efficacy in high-risk populations. Conversely, robust retrospective evidence suggests that in patients with high-risk features-such as advanced T-stage, large tumor size, sarcomatoid differentiation, or venous thrombus-more extensive LND may confer a therapeutic benefit by eradicating micrometastatic disease and improving cancer-specific survival. The advent of effective adjuvant immunotherapy (e.g., pembrolizumab) further underscores the need for accurate nodal staging and re-evaluation of LND's role. This prospective, randomized controlled trial aims to definitively assess the oncological benefit and safety of template-based LND in a rigorously selected high-risk RCC cohort.

Research Objectives:

Primary Objectives:

To compare the impact of RN combined with template lymph node dissection versus RN alone on overall survival (OS) and disease-free survival (DFS) in patients with high-risk RCC.

To evaluate and compare the surgical safety profiles of both approaches, including perioperative complications (graded by Clavien-Dindo classification), operative time, intraoperative blood loss, and length of hospital stay.

Secondary Objectives:

To compare cancer-specific survival (CSS) between the two groups. To quantify the number of lymph nodes retrieved and the incidence of nodal metastases within predefined anatomical templates (renal hilum, para-aortic, paracaval, and interaortocaval regions).

Exploratory Objectives:

To identify molecular biomarkers predictive of nodal metastasis or prognosis using Bulk-RNA sequencing of prospectively collected tumor and blood samples.

To develop a predictive nomogram for lymph node metastasis integrating radiomic features from triple-phase abdominal CT, MRI, tumor characteristics, and clinical symptoms.

Study Methodology:

This is a prospective, open-label, multicenter, randomized controlled trial. A total of 220 eligible patients with high-risk RCC-defined as cT3-4N0-1M0 or M1 disease rendered no evidence of disease (NED) after local therapy-will be randomized in a 1:1 ratio.

Intervention Group (Arm A): Patients will undergo RN plus template LND. The template for left-sided tumors includes lymph nodes from the diaphragmatic crus to the aortic bifurcation (anterior and lateral to the aorta), including the renal hilar nodes. For right-sided tumors, the template extends from the hepatic edge of the inferior vena cava (IVC) to the iliac bifurcation, encompassing paracaval, precaval, and interaortocaval nodes, including the renal hilum.

Control Group (Arm B): Patients will undergo RN with resection only of radiologically or intraoperatively detected lymph nodes ≥1 cm.

Randomization will be centralized and stratified by clinical nodal status (cN0 vs. cN1), prior metastatic status (M0 vs. M1→NED), and participating center. Surgical approach (open, laparoscopic, or robot-assisted) will be at the surgeon's discretion. Postoperative adjuvant therapy with toripalimab (an anti-PD-1 agent) may be offered per patient preference, with one cycle provided free of charge by the study.

Endpoints and Statistical Analysis:

Primary endpoints are DFS and OS. Secondary endpoints include CSS, nodal yield and metastatic rate, and safety. DFS is defined as the time from randomization to recurrence, second primary RCC, or death from any cause. OS is defined as time from randomization to death from any cause. Time-to-event endpoints will be analyzed using Kaplan-Meier methods and compared with the log-rank test. Cox proportional hazards models will be used for multivariable analysis. Categorical variables will be compared using chi-square tests, and continuous variables with t-tests. A sample size of 220 provides 90% power to detect a 21.5% absolute improvement in 5-year OS (76% vs. 54.5%) at a two-sided α of 0.05, accounting for a 10% dropout rate.

Innovation:

This study addresses a critical evidence gap by prospectively evaluating template LND in a meticulously defined high-risk RCC population, including those with M1 NED status-a subgroup with particularly poor prognosis. It employs a standardized, anatomically defined "template" LND to ensure surgical quality and consistency across multiple centers. Furthermore, the study integrates contemporary biomarker and radiomic analyses to explore predictive tools for nodal metastasis and prognosis, which could personalize future surgical and adjuvant strategies. By conducting this trial in the era of adjuvant immunotherapy, it will elucidate whether LND provides independent therapeutic benefit beyond its staging role.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form. Age > 18 years. Candidate for radical nephrectomy with or without lymph node dissection.

High-risk renal cell carcinoma defined as:

At least ONE of: Clinical stage cT3-4 N0-1 M0 (AJCC 8th ed); OR radiologically visible lymph node >1cm; OR M1 disease rendered no evidence of disease (NED) after local therapy; OR radiologically determined rT4 stage.

OR at least TWO of: Renal vein or inferior vena cava tumor thrombus; OR nuclear grade 3-4 or sarcomatoid differentiation or coagulative necrosis; OR tumor size ≥10cm; OR hematuria and/or local symptoms.

Measurable disease as per RECIST v1.1. ECOG performance status of 0 or 1. Adequate bone marrow, renal, and hepatic function. For women and men of childbearing potential, agreement to use effective contraception during the study period.

Exclusion Criteria:

Prior radiotherapy, chemotherapy, major surgery, or targeted therapy for RCC. Concurrent other active malignancy (except controlled malignancies not affecting 2-year survival).

Candidate for partial nephrectomy or ablation per multidisciplinary team assessment.

Preoperative imaging indicates unresectable regional lymph nodes. Bilateral renal tumors or known hereditary RCC syndrome. Diagnosis of any other active malignancy within the past 5 years. Active autoimmune disease or history of autoimmune disease. Use of immunosuppressive agents within 2 weeks prior to enrollment. Poorly controlled cardiac or clinical symptoms. Coagulopathy or bleeding tendency. Active gastrointestinal conditions with risk of bleeding or perforation. History of significant bleeding or thromboembolic events within specified timeframes.

Active infection or unexplained fever >38.5°C. Abdominal fistula, gastrointestinal perforation, or abscess within 4 weeks prior.

History of pulmonary fibrosis, interstitial lung disease, or severely impaired pulmonary function.

Known immunodeficiency or active hepatitis. Participation in another clinical trial within 1 month. Known history of drug abuse or alcohol addiction. Inability or unwillingness to bear the self-paid portion of examination and treatment costs.

Any condition that, in the investigator's judgment, may compromise patient safety or study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From randomization until the first occurrence of disease recurrence, second primary cancer, or death from any cause, assessed up to 10 years.
  Time from randomization to the first documented disease recurrence (local, regional, or distant metastasis), occurrence of a second primary renal cell carcinoma, or death from any cause, whichever occurs first.
Overall Survival (OS) | From randomization until death from any cause, assessed up to 10 years.
  Time from randomization to death from any cause.
Perioperative Safety | From the date of surgery until 30 days post-operation.
  A composite measure to assess the safety of the surgical procedures, including:
  1. Incidence and severity of postoperative complications graded by Clavien-Dindo classification.
  2. Operative time (minutes).
  3. Estimated intraoperative blood loss (milliliters).
  4. Length of postoperative hospital stay (days).

SECONDARY OUTCOMES:
Cancer-Specific Survival (CSS) | From randomization until death from kidney cancer, assessed up to 10 years.
  Time from randomization to death attributable to renal cell carcinoma. Deaths from other causes are censored.
Anatomic Lymph Node Mapping and Metastasis Rate | Assessed on the surgical pathology report, immediately after surgery (within approximately 4 weeks post-operation).
  The absolute number and the pathological nodal positivity rate (pN+%) of lymph nodes retrieved from each of the following predefined anatomical template regions: right renal hilum, suprarenal para-caval, infrarenal para-caval, left renal hilum, suprarenal para-aortic, and renal hilar para-aortic. This assesses the distribution and frequency of lymph node metastasis.
Exploration of Biomarkers for Survival | Biomarker analysis will be conducted after sufficient clinical outcome data (DFS/OS events) are available, estimated to be 5 years after study start.
  Identification of molecular biomarkers predictive of Disease-Free Survival (DFS), Cancer-Specific Survival (CSS), and Overall Survival (OS) through Bulk-RNA sequencing analysis performed on prospectively collected tumor tissue samples.
Predictive Nomogram for Lymph Node Metastasis | Model development and internal validation will be performed after complete recruitment and surgical pathology data are available for all participants, estimated to be 3 years after study start.
  Development and validation of a predictive nomogram (statistical model) for preoperative estimation of lymph node metastasis risk. The model will integrate radiomic features from contrast-enhanced abdominal CT and non-contrast MRI, along with clinical variables (tumor size/location, retroperitoneal/renal hilar lymph node size/location, and clinical symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Quan, MD, Principal Investigator — Tianjin Medical University Second Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] Capitanio U, Matloob R, Suardi N, Abdollah F, Castiglione F, Di Trapani D, Russo A, Briganti A, Carenzi C, Salonia A, Montorsi F, Rigatti P, Bertini R. The extent of lymphadenectomy does affect cancer specific survival in pathologically confirmed T4 renal cell carcinoma. Urologia. 2012 Apr-Jun;79(2):109-15. doi: 10.5301/RU.2012.9255. PMID 22610843
- [Background] Capitanio U, Suardi N, Matloob R, Roscigno M, Abdollah F, Di Trapani E, Moschini M, Gallina A, Salonia A, Briganti A, Montorsi F, Bertini R. Extent of lymph node dissection at nephrectomy affects cancer-specific survival and metastatic progression in specific sub-categories of patients with renal cell carcinoma (RCC). BJU Int. 2014 Aug;114(2):210-5. doi: 10.1111/bju.12508. Epub 2014 May 22. PMID 24854206
- [Background] Whitson JM, Harris CR, Reese AC, Meng MV. Lymphadenectomy improves survival of patients with renal cell carcinoma and nodal metastases. J Urol. 2011 May;185(5):1615-20. doi: 10.1016/j.juro.2010.12.053. Epub 2011 Mar 21. PMID 21419453
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Crispen PL, Breau RH, Allmer C, Lohse CM, Cheville JC, Leibovich BC, Blute ML. Lymph node dissection at the time of radical nephrectomy for high-risk clear cell renal cell carcinoma: indications and recommendations for surgical templates. Eur Urol. 2011 Jan;59(1):18-23. doi: 10.1016/j.eururo.2010.08.042. Epub 2010 Sep 15. PMID 20933322
- [Background] Motzer RJ, Jonasch E, Agarwal N, Alva A, Baine M, Beckermann K, Carlo MI, Choueiri TK, Costello BA, Derweesh IH, Desai A, Ged Y, George S, Gore JL, Haas N, Hancock SL, Kapur P, Kyriakopoulos C, Lam ET, Lara PN, Lau C, Lewis B, Madoff DC, Manley B, Michaelson MD, Mortazavi A, Nandagopal L, Plimack ER, Ponsky L, Ramalingam S, Shuch B, Smith ZL, Sosman J, Dwyer MA, Gurski LA, Motter A. Kidney Cancer, Version 3.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Jan;20(1):71-90. doi: 10.6004/jnccn.2022.0001. PMID 34991070
- [Background] Hutterer GC, Patard JJ, Perrotte P, Ionescu C, de La Taille A, Salomon L, Verhoest G, Tostain J, Cindolo L, Ficarra V, Artibani W, Schips L, Zigeuner R, Mulders PF, Valeri A, Chautard D, Descotes JL, Rambeaud JJ, Mejean A, Karakiewicz PI. Patients with renal cell carcinoma nodal metastases can be accurately identified: external validation of a new nomogram. Int J Cancer. 2007 Dec 1;121(11):2556-61. doi: 10.1002/ijc.23010. PMID 17691107
- [Background] Babaian KN, Kim DY, Kenney PA, Wood CG Jr, Wong J, Sanchez C, Fang JE, Gerber JA, Didic A, Wahab A, Golla V, Torres C, Tamboli P, Qiao W, Matin SF, Wood CG, Karam JA. Preoperative predictors of pathological lymph node metastasis in patients with renal cell carcinoma undergoing retroperitoneal lymph node dissection. J Urol. 2015 Apr;193(4):1101-7. doi: 10.1016/j.juro.2014.10.096. Epub 2014 Oct 25. PMID 25390078
- [Background] Choueiri TK, Tomczak P, Park SH, Venugopal B, Ferguson T, Symeonides SN, Hajek J, Chang YH, Lee JL, Sarwar N, Haas NB, Gurney H, Sawrycki P, Mahave M, Gross-Goupil M, Zhang T, Burke JM, Doshi G, Melichar B, Kopyltsov E, Alva A, Oudard S, Topart D, Hammers H, Kitamura H, McDermott DF, Silva A, Winquist E, Cornell J, Elfiky A, Burgents JE, Perini RF, Powles T; KEYNOTE-564 Investigators. Overall Survival with Adjuvant Pembrolizumab in Renal-Cell Carcinoma. N Engl J Med. 2024 Apr 18;390(15):1359-1371. doi: 10.1056/NEJMoa2312695. PMID 38631003
- [Background] Margulis V, Wood CG. The role of lymph node dissection in renal cell carcinoma: the pendulum swings back. Cancer J. 2008 Sep-Oct;14(5):308-14. doi: 10.1097/PPO.0b013e31818675eb. PMID 18836335
- [Background] Gershman B, Moreira DM, Thompson RH, Boorjian SA, Lohse CM, Costello BA, Cheville JC, Leibovich BC. Perioperative Morbidity of Lymph Node Dissection for Renal Cell Carcinoma: A Propensity Score-based Analysis. Eur Urol. 2018 Mar;73(3):469-475. doi: 10.1016/j.eururo.2017.10.020. Epub 2017 Nov 11. PMID 29132713
- [Background] Bex A, Ghanem YA, Albiges L, Bonn S, Campi R, Capitanio U, Dabestani S, Hora M, Klatte T, Kuusk T, Lund L, Marconi L, Palumbo C, Pignot G, Powles T, Schouten N, Tran M, Volpe A, Bedke J. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2025 Update. Eur Urol. 2025 Jun;87(6):683-696. doi: 10.1016/j.eururo.2025.02.020. Epub 2025 Mar 20. PMID 40118739
- [Background] Pantuck AJ, Zisman A, Dorey F, Chao DH, Han KR, Said J, Gitlitz BJ, Figlin RA, Belldegrun AS. Renal cell carcinoma with retroperitoneal lymph nodes: role of lymph node dissection. J Urol. 2003 Jun;169(6):2076-83. doi: 10.1097/01.ju.0000066130.27119.1c. PMID 12771723
- [Background] Gershman B, Thompson RH, Moreira DM, Boorjian SA, Tollefson MK, Lohse CM, Costello BA, Cheville JC, Leibovich BC. Radical Nephrectomy With or Without Lymph Node Dissection for Nonmetastatic Renal Cell Carcinoma: A Propensity Score-based Analysis. Eur Urol. 2017 Apr;71(4):560-567. doi: 10.1016/j.eururo.2016.09.019. Epub 2016 Sep 24. PMID 27671144
- [Background] Zi H, Liu MY, Luo LS, Huang Q, Luo PC, Luan HH, Huang J, Wang DQ, Wang YB, Zhang YY, Yu RP, Li YT, Zheng H, Liu TZ, Fan Y, Zeng XT. Global burden of benign prostatic hyperplasia, urinary tract infections, urolithiasis, bladder cancer, kidney cancer, and prostate cancer from 1990 to 2021. Mil Med Res. 2024 Sep 18;11(1):64. doi: 10.1186/s40779-024-00569-w. PMID 39294748
- [Background] Blom JH, van Poppel H, Marechal JM, Jacqmin D, Schroder FH, de Prijck L, Sylvester R; EORTC Genitourinary Tract Cancer Group. Radical nephrectomy with and without lymph-node dissection: final results of European Organization for Research and Treatment of Cancer (EORTC) randomized phase 3 trial 30881. Eur Urol. 2009 Jan;55(1):28-34. doi: 10.1016/j.eururo.2008.09.052. Epub 2008 Oct 1. PMID 18848382
- [Background] Capitanio U, Becker F, Blute ML, Mulders P, Patard JJ, Russo P, Studer UE, Van Poppel H. Lymph node dissection in renal cell carcinoma. Eur Urol. 2011 Dec;60(6):1212-20. doi: 10.1016/j.eururo.2011.09.003. Epub 2011 Sep 13. PMID 21940096
- [Background] Ngai M, Chandrasekar T, Bratslavsky G, Goldberg H. The Current Role of Lymph Node Dissection in Nonmetastatic Localized Renal Cell Carcinoma. J Clin Med. 2023 May 29;12(11):3732. doi: 10.3390/jcm12113732. PMID 37297925
- [Background] Marshall FF, Powell KC. Lymphadenectomy for renal cell carcinoma: anatomical and therapeutic considerations. J Urol. 1982 Oct;128(4):677-81. doi: 10.1016/s0022-5347(17)53132-8. No abstract available. PMID 7143582
- [Background] Blute ML, Leibovich BC, Cheville JC, Lohse CM, Zincke H. A protocol for performing extended lymph node dissection using primary tumor pathological features for patients treated with radical nephrectomy for clear cell renal cell carcinoma. J Urol. 2004 Aug;172(2):465-9. doi: 10.1097/01.ju.0000129815.91927.85. PMID 15247704
- [Background] Capitanio U, Leibovich BC. The rationale and the role of lymph node dissection in renal cell carcinoma. World J Urol. 2017 Apr;35(4):497-506. doi: 10.1007/s00345-016-1886-3. Epub 2016 Jun 30. PMID 27364520

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT07321197/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT07321197/ICF_001.pdf